CLINICAL TRIAL: NCT06064006
Title: A Randomised, Placebo-controlled and Double-blinded Study Assessing the Safety, Tolerability, Pharmacokinetics, and Efficacy of Subcutaneous Administrations of NNC0487-0111 in Participants With Overweight or Obesity
Brief Title: A Research Study to See How a New Medicine (NNC0487-0111) Works in People With Overweight or Obesity When Injected Under the Skin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9490-7613; U1111-1289-3282 (Other: World Health Organization (WHO))
Record Dates: First submitted 2023-09-11; First posted 2023-10-03 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NNC0487-0111 (Experimental): Participants will be randomized to receive NNC0487-0111. The study will be conducted in 5 parts. Part A: Single ascending dose (SAD) Part B, C, D and E: Multiple ascending dose (MAD)
  Interventions: Drug: NNC0487-0111; Drug: Placebo (NNC0487-0111)
- Placebo (Placebo Comparator): Participants will be randomized to receive Placebo. The study will be conducted in 5 parts. Part A: Single ascending dose (SAD). Part B,C,D and E: Multiple ascending dose (MAD).
  Interventions: Drug: NNC0487-0111; Drug: Placebo (NNC0487-0111)

INTERVENTIONS:
Drug: NNC0487-0111 — NNC0487-0111 will be administered as a subcutaneous (s.c. under the skin) injection.
Drug: Placebo (NNC0487-0111) — Placebo matching NNC0487-0111 will be administered as a subcutaneous (s.c. under the skin) injection.

SUMMARY:
The purpose of the study is to evaluate if a new study drug, NNC0487-0111, is safe and how it works in the participant's body, when given as injections under the skin

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Aged 18-55 years (both inclusive) at the time of signing informed consent.
* Body Mass Index (BMI) between 27.0 and 39.9 kg/m^2 (both inclusive) at screening. Overweight should be due to excess adipose tissue, as judged by the investigator.
* Considered eligible based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests performed during the screening visit, as judged by the investigator.

Exclusion Criteria:

* Any disorder, which in the investigator's opinion might jeopardise participant's safety or compliance with the protocol
* HbA1c equal to or greater than 6.5 % (48 mmol/mol) at screening
* Any laboratory safety parameters at screening outside the below laboratory ranges, see designated reference range documents for specific values:

  * Vitamin D (25-hydroxycholecalciferol) below 12 ng/mL (30 nM) at screening
  * Parathyroid hormone (PTH) outside normal range at screening
  * Total calcium outside normal range at screening
  * Amylase equal to or greater than 2 times upper limit of normal at screening
  * Lipase equal to or greater than 2 times upper limit of normal at screening
  * Calcitonin equal to or greater than 50 ng/L at screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 125 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-11-27 (Actual); Study Completion 2024-11-27 (Actual)

PRIMARY OUTCOMES:
PART A: Number of treatment emergent adverse events (TEAE) | From pre-dose on Day 1 until completion of the end of study visit, up to Day 25
  Number of events
PARTS B to E: Number of treatment emergent adverse events (TEAE) | From pre-dose on Day 1 until completion of the end of study visit (V37) up to Day 270
  Number of events

SECONDARY OUTCOMES:
PART A: AUC0-∞,SD; the area under the NNC0487-0111 plasma concentration-time curve from time 0 to infinity after a single dose | From pre-dose on Day 1 until completion of the end of study visit, up to Day 25
  h*nmol/L
PART A: Cmax,SD; the maximum plasma concentration of NNC0487-0111 after a single dose and the corresponding time tmax | From pre-dose on Day 1 until completion of the end of study visit, up to Day 25
  nmol/L
PARTS B to E: AUC0-168h,SS; the area under the NNC0487-0111 plasma concentration-time curve from time 0 to 168 hours after last multiple dose | From pre-dose on V33D1 until end of treatment (V34) up to 9 days
  h*nmol/L
PARTS B to E: Cmax,SS; the maximum plasma concentration of NNC0487-0111 after last multiple dose and the corresponding time tmax | From pre-dose on V33D1 until end of study visit (V37) up to 24 days
  nmol/L
PART B to E: Relative change in body weight | From pre-dose on Day 1 until end of treatment (V34) up to Day 255
  Percentage (%)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency dept. 2834, Study Director — Novo Nordisk A/S
Locations (2):
- United States (2):
  - ICON Early Phase Services, LLC, San Antonio, Texas
  - Novo Nordisk INvestigational Site, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com.
URL: http://novonordisk-trials.com

REFERENCES:
- [Derived] Dahl K, Toubro S, Dey S, Duque do Vale R, Flint A, Gasiorek A, Heydorn A, Jastreboff AM, Key C, Petersen SB, Vegge A, Adelborg K. Amycretin, a novel, unimolecular GLP-1 and amylin receptor agonist administered subcutaneously: results from a phase 1b/2a randomised controlled study. Lancet. 2025 Jul 12;406(10499):149-162. doi: 10.1016/S0140-6736(25)01185-7. Epub 2025 Jun 20. PMID 40550231